CLINICAL TRIAL: NCT06537609
Title: BALANCE+: A Platform Trial for Gram Negative Bloodstream Infections
Brief Title: A Platform Trial for Gram Negative Bloodstream Infections
Acronym: BALANCE+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Clínica Universidad de La Sabana (Unknown); Universidad de La Sabana, Colombia (Unknown); Aotearoa Clinical Trials (Unknown)
Responsible Party: Principal Investigator, Dr. Nick Daneman, Clinician Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4369-1
Record Dates: First submitted 2024-07-25; First posted 2024-08-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: Gram-negative Bacteremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- De-escalation VS No De-escalation (Active Comparator)
  Interventions: Other: De-escalation VS No De-escalation
- Oral beta-lactams VS Oral Non-beta-lactams (Active Comparator)
  Interventions: Other: Oral beta-lactams VS non beta-lactams
- Central vascular catheter retention VS Central vascular catheter replacement (Active Comparator)
  Interventions: Other: Central vascular catheter retention VS Central vascular catheter replacement
- Cephalosporin VS Carbapenem for low risk AmpC organisms (Active Comparator)
  Interventions: Other: Cephalosporin VS Carbapenem for low risk AmpC organisms
- Routine follow-up blood culture VS No routine follow-up blood culture (Active Comparator)
  Interventions: Other: Routine follow-up blood culture VS No routine follow-up blood culture

INTERVENTIONS:
Other: De-escalation VS No De-escalation — No de-escalation group: continue to receive the same antibiotic that was started initially (as long as it is confirmed to be effective based on the blood culture sensitivity result). De-escalation is only allowed within 7 days if patient is being discharged from hospital.
  De-escalation group: switched to narrower spectrum antibiotic (based on spectrum scale specified in protocol).
  Arms: De-escalation VS No De-escalation
Other: Oral beta-lactams VS non beta-lactams — Beta-lactam antibiotic: This can be, but not limited to, amoxicillin, amoxicillin-clavulanate, cephalexin, cefadroxil, or cefixime.
  Non beta-lactam antibiotic: This can be ciprofloxacin, moxifloxacin, levofloxacin or trimethoprim-sulfamethoxazole.
  Arms: Oral beta-lactams VS Oral Non-beta-lactams
Other: Central vascular catheter retention VS Central vascular catheter replacement — Central vascular catheter replacement: the catheter will be changed by the treating team as soon as possible and within a maximum of 72 hours from blood culture finalization
  Central vascular catheter retention: the catheter will not be changed and will be retained until it is non functional or no longer needed.
  Arms: Central vascular catheter retention VS Central vascular catheter replacement
Other: Cephalosporin VS Carbapenem for low risk AmpC organisms — Cephalosporin (ceftriaxone) at standard doses
  Carbapenem (Meropenem or Ertapenem) at standard doses
  Arms: Cephalosporin VS Carbapenem for low risk AmpC organisms
Other: Routine follow-up blood culture VS No routine follow-up blood culture — Routine follow-up blood culture: routine repeat blood collection 4 days from the index blood collection with positive bacteria.
  No follow-up blood culture: no routine repeat blood collection 4 days from the index blood collection with positive bacteria
  Arms: Routine follow-up blood culture VS No routine follow-up blood culture

SUMMARY:
BALANCE+ is a perpetual multiple domain randomized controlled platform trial to evaluate various treatment strategies for Gram-negative bloodstream infections (GN BSIs). Each domain addresses critical questions in the management of GN BSIs, aiming to refine treatment strategies, enhance patient outcomes, and reduce antimicrobial resistance.

The initial vanguard pilot RCT (NCT05893147) started on 29 August 2023 and has successfully completed the pilot phase on 24-Apr-2024. All patients enrolled in the vanguard phase are part of the main platform trial.

DETAILED DESCRIPTION:
BALANCE+ is an adaptive platform trial evaluating multiple treatment options in patients admitted to the hospital due to Gram negative bloodstream infections (BSIs). It focuses on both cross-cutting and subgroup-specific questions, using an open-label, pragmatic design embedded in routine care.

BALANCE+ addresses the significant health concern of BSIs, which have high morbidity and mortality rates, exacerbated by the global public health threat of antimicrobial resistance (AMR). With rising resistance rates and limited new drug development, effective treatment strategies for BSIs remain under-researched.

BALANCE+ follows the BALANCE trial, which evaluated duration of antibiotic treatment, and aims to further investigate critical questions in managing Gram-negative BSIs. This platform trial will explore various aspects of BSI treatment, including antibiotic de-escalation, oral antibiotic choices, central line management, treatment of specific pathogens, and the necessity of follow-up blood cultures.

BALANCE+ is using Bayesian methods without a fixed sample size. Interim analyses will occur after every 1000th patient in each domain, and then for every 200th patient thereafter. The trial will stop if futility or superiority thresholds are met, or if a domain reaches its ceiling sample size (2500 patients for most domains and 4000 for the beta-lactam versus non-beta-lactam domain) without meeting a stopping threshold.

A vanguard pilot trial involving over 150 patients at 9 hospitals across Canada confirmed the feasibility of the BALANCE+ trial. The main trial will include patients from the vanguard pilot phase since there has been no major change in the overall study design and domains. The adaptive design allows for interim analyses and adjustments by adding or removing domains as per the statistical analysis plan, enhancing the trial's efficiency and relevance.

ELIGIBILITY:
PLATFORM INCLUSION CRITERIA

Platform Inclusion Criteria:

* admitted to a participating hospital
* positive blood culture with Gram negative (GN) bacterium

Platform Exclusion Criteria:

* patient's goals of care are for palliation with no active treatment
* moribund patient, not expected to survive > 72 hours
* previously enrolled in the platform trial
* not eligible for any domain at the time of screening

DOMAIN SPECIFIC INCLUSION AND EXCLUSION CRITERIA

1. De-escalation versus no de-escalation domain

   Inclusion Criteria

   - included in BALANCE+ platform

   Exclusion Criteria
   * receiving an empiric antibiotic regimen at the time of blood culture finalization to which the GN pathogen(s) are not sensitive
   * arbapenem-non-susceptible
   * no de-escalation option due to any or all of:

     * antimicrobial resistance
     * allergies
     * medical contraindications
     * drug-drug interaction risk
     * other relevant reason
   * patients with a suspected or proven polymicrobial source of infection
   * > 24 hours since index blood culture susceptibility results finalization
2. Beta-lactam versus non-beta-lactam oral/enteral treatment domain

   Inclusion Criteria
   * included in BALANCE+ platform
   * initially treated with intravenous antibiotics, but clinical team transitioning patient to oral/enteral antibiotic within 7 days of starting treatment

   Exclusion Criteria
   * enrolled in an arm of another BALANCE+ platform domain which limits the use of oral/enteral therapy:
   * no-de-escalation arm (patients in the no de-escalation arm cannot be randomized into this domain unless they are ready for discharge home, in which case de-escalation is allowable to oral agents at discharge)
   * no non-beta-lactam options due to any or all of:

     * resistance
     * allergies
     * medical contraindications
     * drug-interaction risk
     * other relevant reason
   * no beta-lactam options due to any or all of:

     * resistance
     * allergies
     * medical contraindications
     * drug-interaction risk
     * other relevant reason
   * pregnancy
   * already received >24 hours of oral antibiotics after index blood culture finalization
3. Central vascular catheter replacement domain

   Inclusion Criteria
   * included in BALANCE+ platform
   * has an indwelling central vascular catheter that was already in place within the 48-hour period before the onset of bloodstream infection (i.e. is not a new catheter placed within 48 hours of the onset of infection)

   Exclusion Criteria
   * patient has no ongoing need for a central vascular catheter
   * patient has definite indication for central vascular catheter removal
   * ongoing septic shock with definite/probable line source

     * concomitant S. aureus bacteremia
     * concomitant candidemia
   * local suppurative signs (severe redness, warmth, pain, swelling or fluctuance/collection) necessitating catheter removal, or other clinical evidence of infected line (e.g. imaging/echocardiographic findings)
4. Low-risk AmpC domain

   Inclusion Criteria
   * included in BALANCE+ platform
   * positive blood culture with GN bacterium, of the following species: i. Serratia spp. ii Morganella spp. iii Providencia spp. iv Proteus spp. other than P.mirabilis
   * organism is susceptible to ceftriaxone

   Exclusion Criteria
   * severe allergy to beta-lactams (e.g., type 4 hypersensitivity reaction or DRESS)
   * baseline phenotypic non-susceptiblity to ceftriaxone
   * more than 1 calendar day beyond availability of susceptibility results
5. Follow up blood culture domain

Inclusion Criteria

- included in BALANCE+ platform

Exclusion Criteria

* patient died or discharged from hospital prior to day 4
* blood culture already collected by the treating team at day 4±1
* >5 days since index positive blood culture collection
* definite indication for repeat blood culture testing

  * concomitant S. aureus bacteremia
  * concomitant Candidemia
  * clinical suspicion for infective endocarditis

Ages: 0 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Desirability of Outcome Ranking (DOOR) Ordinal Scale which incorporates death, reinfection, readmission, and for some domains incorporates a tie-breaker of new antimicrobial resistance (AMR). | 90 days
  The primary outcome for each domain will use a Desirability of Outcome Ranking (DOOR) ordinal scale in which patients are categorized into the following mutually exclusive categories, ranked from best to worst status:
  1. Alive with no reinfection or readmission.
  2. Alive with reinfection OR readmission.
  3. Alive with reinfection AND readmission.
  4. Dead
  For the 3 antibiotic-related domains (the de-escalation versus no de-escalation domain, the beta-lactam versus non-beta-lactam domain, and the low risk AmpC domain) there will be an additional tie-breaker within ordinal levels 1, 2 and 3 based on whether there was new detection of antimicrobial resistance (AMR).

SECONDARY OUTCOMES:
90-day mortality | 90 days
90-day re-infection | 90 days
90-day all cause readmission | 90 days
90-day AMR colonization/infection | 90 days
90-day Clostridioides difficile infection (CDI) | 90 days
30-day mortality | 30 days
60-day mortality | 60 days
Additional Secondary Outcomes for Individual Domains | 90 days
  (i) De-escalation versus no de-escalation
  * change in total microbiome diversity between the day of randomization and discharge (or day 30 if earlier)
  * net change in resistome AMR burden between the day of randomization and discharge (or day 30 if earlier).
  (ii) Beta-lactam versus non-beta-lactam
  * antibiotic-related allergic reaction
  * antibiotic-related adverse event
  (iii) Central vascular catheter replacement versus retention
  * pneumothorax or thoracotomy tube insertion related to vascular catheter
  * clinically important bleeding
  * line associated thrombus
  * persistent bacteremia >5d from initial index culture
  * secondary bloodstream infection with new bacterial or fungal organism
  (iv) Low-risk AmpC
  * isolation of ESBL producing organism or third generation cephalosporin resistant Gram negative organism
  * isolation of a carbapenem-resistant organism
    (v) Follow up blood culture domain
  * total duration of antibiotic therapy
  * hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Nick Daneman, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Rob Fowler, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (39):
- Australia (8):
  - St George Hospital, Kogarah, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Sunshine Coast University Hospital, Sunshine Coast, Queensland
  - Monash Medical Center, Clayton, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - St John of God, Murdoch, Western Australia
- Canada (28):
  - Foothills Hospital, Calgary, Alberta
  - Peter Lougheed Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Grace Hospital, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Dr. Everett Chalmers Regional Hospital, Fredericton, New Brunswick
  - Eastern Regional Health Authority, St. John's, Newfoundland and Labrador
  - Trillium Health Partners - Mississauga Hospital, Mississauga, Ontario
  - Humber River Health system, North York, Ontario
  - North York General Hospital, North York, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CHU de Québec - Université Laval, Laval, Quebec
  - Hôpital de la Cité de la Santé, Laval, Quebec
  - Montreal General Hospital- McGill, Montreal, Quebec
  - Royal Victoria Hospital- McGill, Montreal, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec
  - Centre hospitalier affilié universitaire régional (CHAUR), Trois-Rivières, Quebec
- Universidad de La Sabana, Chía, Cundinamarca, Colombia
- Sheba Medical Center, Ramat Gan, Tel Aviv, Israel
- Middlemore Hospital, Auckland, Auckland, New Zealand